CLINICAL TRIAL: NCT06311084
Title: IMAGINATOR 2.0: Co-design and Early Evaluation of a Novel Blended Digital Intervention Targeting Self-harm in Young People
Acronym: IMAG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 310211
Record Dates: First submitted 2024-02-19; First posted 2024-03-15 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Self Injurious Behavior; Adolescent Behavior Problem; Child Behavior Problem; Mental Health Disorder
Keywords: Self Injurious Behaviour; Mental Health Disorder
MeSH Terms: conditions — Self-Injurious Behavior; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Open ended feasibility and acceptability of novel blended digital psychological intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginator - Functional Imagery Training (Experimental): 3 weekly face to face sessions of Functional Imagery Training, followed by 5 fortnightly phone support calls, and the Imaginator app
  Interventions: Other: Imaginator 2.0

INTERVENTIONS:
Other: Imaginator 2.0 — Blended psychological digital intervention, combining Functional Imagery Training, a psychological intervention based on CBT and motivational interviewing principles, and a smartphone app.

SUMMARY:
This study aims to investigate acceptability and feasibility of a new version of the Imaginator intervention, Imaginator 2.0, targeting self-harm behaviour in young people aged 12-25 under mental health services in the UK.

Following an initial proof-of-concept study of Imaginator (Di Simplicio et al., 2020), a new version of the app that supports consolidation and practice of the techniques learnt in therapy was co-designed, and the protocol was adapted to be extended to younger adolescents.

Imaginator 2.0 uses 'functional imagery training', training in individuals to develop and use functional (that is, helpful) mental images to support an alternative behaviour instead of self-harm. Mental imagery is the process of picturing something in the mind, and mental images have strong emotional and motivational characteristics. Functional Imagery Training (FIT) within Imaginator helps young people imagine adaptive behaviours as an alternative to self-harm when dealing with distressing emotions.

DETAILED DESCRIPTION:
An open single-arm study that investigates the IMAGINATOR intervention comprising of delivery of Functional Imagery Training (FIT) for self-harm supported by a new co-designed smartphone app for young people aged 12-25 who experience current repeated self-harming behaviour and have been referred to adult community mental health services (Mental Health Integrated Network Teams; MINT) or Community Child and Adolescent Mental Health Services (CAMHS).

For the purpose of this study, self-harm is defined as per NICE guidelines (NICE, 2012): "an act of self-poisoning or self-injury, irrespective of the apparent purpose of the act".

The IMAGINATOR intervention has been tested with 16-25 year olds using a proof of concept trial (Di Simplicio et al., 2020) but as the current study proposes to also include younger participants (12-17 year olds) and a newly co-produced version of the IMAGINATOR app, an open single-arm trial is the optimal design to assess the feasibility and acceptability of the new IMAGINATOR intervention following further protocol/materials development and with a different population.

The IMAGINATOR intervention provides three face-to-face sessions of FIT, followed by phone support sessions and smartphone app-based support, based on cognitive behavioural and motivational interviewing principles and in line with NICE guidelines for long-term management of self-harm behaviour. FIT is intended as a brief and focused transdiagnostic intervention that can be added to any other pharmacological or non-concurrent psychological therapy. To improve YP's access to and engagement with the intervention, FIT was combined with the new IMAGINATOR smartphone app.

The study is based in the West London NHS Trust.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12 - 25 years old
2. Presented with at least 2 episodes of self-harm lifetime, with at least 1 of these in the past month or 5 episodes of self-harm in the past year (based on NSSI Disorder criteria in the DSM-5) and currently reporting self-harm urges or difficulties stopping
3. Have a smartphone
4. Can commit to attending 3 consecutive weekly FIT sessions, and 5 follow-up telephone sessions, and assessments over follow up period as required by the study
5. Have adequate English language ability to permit the assessment and experimental measures to be completed, and use the smartphone app
6. Willing to consent to receive support to reduce / improve management of self-harm urges and behaviour; in person or by video, and over the phone and via smartphone app
7. If 12 - 15 years old, willing for parent/guardian to provide consent to study participation
8. Willing to have letters sent/phone calls made to their GP and other relevant clinicians
9. Resident within geographical areas covered by the West London NHS Trust CCAMHS and MINT teams.

Exclusion Criteria:

The participant may not enter the study if any of the following apply:

1. Severe learning disability or pervasive developmental disorder
2. Current acute psychotic episode
3. Current substance dependence
4. Imminent risk of suicide or harm to others (based on clinicians' risk assessment, see Section 4.1)
5. Insufficient English language fluency to complete study outcome measures
6. Taking part in concurrent treatment studies investigating pharmacological or psychological treatment for self-harm
7. Unwilling to engage actively in the FIT intervention or to use an imagery-focused approach for treatment
8. Unwilling to use a smartphone app.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West London NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Di Simplicio M, Appiah-Kusi E, Wilkinson P, Watson P, Meiser-Stedman C, Kavanagh DJ, Holmes EA. Imaginator: A Proof-of-Concept Feasibility Trial of a Brief Imagery-Based Psychological Intervention for Young People Who Self-Harm. Suicide Life Threat Behav. 2020 Jun;50(3):724-740. doi: 10.1111/sltb.12620. Epub 2020 Feb 14. PMID 32057131
- [Derived] Servi A, Gardner-Bougaard E, Mohamed S, McDermott A, Rodrigues R, Aveyard B, Van Zalk N, Hampshire A, Dewa L, Di Simplicio M. Early Evaluation of IMAGINATOR 2.0 Intervention Targeting Self-Harm in Young People: Single-Arm Feasibility Trial. JMIR Form Res. 2026 Jan 26;10:e79496. doi: 10.2196/79496. PMID 41587082

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol initially planned for the enrolment of 20 participants, with the aim of analysing data from 15 participants who completed the study. However, we received more referrals than anticipated and 29 were eligible and analysed to account for potential attrition and ultimately, 15 participants completed the study, aligning with our target for analysis.
Groups:
- Imaginator App Plus Therapy: After Baseline screening visit, participants received 3 x 1-hour Functional Imagery Training (FIT) sessions in person or via MS Teams once a week. Therapy sessions were delivered by a Child Wellbeing Practitioner (CWP), Clinical Assistant Psychology Therapists (CAPT) or therapist. After completion of the 3 therapy sessions, participants received 5 x 15-30-minute phone-call support sessions fortnightly. FIT comprised of the following key elements: Session 1 - formulation of personal drivers of SH behaviour and motivational interviewing combined with mental imagery techniques; Session 2 - mental imagery of a past achievement, formulation of goals (e.g.,a desired behaviour incompatible with or alternative to SH) and functional imagery plan to achieve them; Session 3 - practice and refinement of functional imagery, problem-solving of challenges. Follow-up phone-call sessions focused on refining functional imagery practice, problem-solving, motivational encouragement, and personalisation of the app use. Participants receiveed smartphone app-based reminders (from Imaginator app), exercises and support from the second FIT session. Upon completion of the follow-up sessions, participants were invited to an outcome assessment after 1 week, at approximately 3 months post intervention. Optional user-led feedback interviews with participants were carried out upon study completion (after final assessment).
Period: Overall Study
Arm/Group | Imaginator App Plus Therapy
Started | 29
Completed | 15
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.86 (3.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 28
  Transgender | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17
  Black, African, Caribbean or Black British | 4
  Mixed or Multiple ethnic groups | 3
  Asian of Asian British | 2
  Other ethnic group | 3
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 12
  Other | 12
  Homosexual | 3
  Not sure | 2
Highest level of education completed [Count of Participants; unit: Participants]
  Postgraduate education | 1
  Higher education | 7
  Secondary education | 13
  Primary education | 8
Household Income [Count of Participants; unit: Participants]
  <50,000 | 18
  50,000 - 100,000 | 9
  100,000 - 150,000 | 1
  150,000 - 200,000 | 1
Currently in education training [Count of Participants; unit: Participants]
  Yes | 14
  No | 15
Employment status [Count of Participants; unit: Participants]
  Yes - Employed | 14
  No - Not Employed | 15
Timeline Follow-Back Technique (TLFB) [Median (Inter-Quartile Range); unit: units on a scale] — This is an interview method conducted by the researcher who reconstructs together with the participant the number of self-harm behaviours using calendar cues. The scale records the total number of self-harm episodes within a specified timeframe of the last 3 months, with higher values indicating more frequent self-harm behaviours. The minimum number of episodes is 0 and the maximum number of episodes that can be reported for the 3 months is every day (so around 90 depending on the number of days of the month). Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 7.5 [5.25 to 26]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 6.5 [3.25 to 28.25]
Self-Harm Imagery Interview (PANAS+) [Median (Inter-Quartile Range); unit: units on a scale] — PANAS+ assesses positive emotions about mental images that deal with self-harm/ occur with self-harm. It is a 10-item scale with items rated on a 5-point Likert scale ranging from 1 (very low intensity or absence of specific emotion) to 5 (extremely high intensity of that emotion). Total scores range from 10 reflecting low positive emotional intensity (weak or minimal positive emotions associated with imagery), to 50 reflecting high positive emotional intensity (strong and vivid positive emotions). Higher scores indicate a greater intensity of positive emotional experiences related to imagery. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 16 [13.5 to 22]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 14 [13 to 22]
Self-Harm Imagery Interview (PANAS-) [Median (Inter-Quartile Range); unit: units on a scale] — PANASi assesses negative emotions about mental images that deal with self-harm/ occur with self-harm. It is a 10-item scale with items rated on a 5-point Likert scale ranging from 1 (very low intensity or absence of specific emotion) to 5 (extremely high intensity of that emotion). Total scores range from 10 reflecting low negative emotional intensity (weak or minimal positive emotions associated with imagery), to 50 reflecting high negative emotional intensity (strong and vivid positive emotions). Higher scores indicate a greater intensity of negative emotional experiences related to imagery. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 32 [24.5 to 41]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 33 [29.5 to 41]
State Motivation for Reducing Self-harm (SM-SH) scale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 12 item scale measures motivation to control self-harm. Each item is rated on a 10-point Likert scale ranging from 0 (never), indicating that the participant has no motivation or desire to control their self-harm, to 10 (constantly), indicating that the participant has an extremely strong and persistent motivation to control their self-harm. Average scores are calculated for each participant ranging from 0 to 10, with higher scores indicating stronger motivation to control self-harm. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 5.67 [4.38 to 7.02]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 5.33 [4.62 to 6.36]
Craving Experience Questionnaire for Self-Harm (CEQ-SH) [Median (Inter-Quartile Range); unit: units on a scale] — This 9-item measure assesses the urge to self-harm and frequency, intensity, salience or dismissability of intrusive thoughts surrounding self-harm. Each item is rated on a 10-point Likert scale ranging from 0 (not at all), indicating no urge to self-harm or does not experience any intrusive thoughts related to self-harm, to 10 (constantly), indicating a very strong and persistent urge to self-harm or constantly preoccupied with thoughts of self-harm. The minimum score is 0, indicating no urge to self-harm, and the maximum score is 90, indicating the highest possible urge to self-harm. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 60 [44.75 to 70]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 59 [43.5 to 67.5]
Revised Children's Anxiety and Depression Scale (RCADS) - Anxiety subscale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 47 item measure for 12-17 year olds. This analysis focuses on the Anxiety sub-scales (37 items). Each item is scored from 0 (never), indicating not experiencing the symptom described in the item during the past week, to 3 (always), consistently experiencing the symptom. Total scores range from 0 to 111. A total score is calculated by summing the individual item scores. Higher scores indicate more severe anxiety. Here raw scores are reported. Population: This measure is only for 12-17 year olds, so only people in this age range are analysed. Initially, we enrolled 29 participants out of which 11 were 12-17 years old (analysed in first row). As we were interested in changes before and after the intervention, we also report the baseline results just for the participants who completed the outcome assessment. Out of the 15 participants who completed the outcome assessment, 7 were 12-17 years old (analysed in second row).
  units on a scale
    All Baseline Participants: number analyzed (Participants) | 11
    All Baseline Participants | 68 [49 to 72]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 7
    Participants who completed the Outcome Assessment | 57 [38.5 to 67.5]
Revised Children's Anxiety and Depression Scale (RCADS) - Depression subscale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 47 item measure for 12-17 year olds. This analysis focuses on the Depression sub-scale (10 items). Each item is scored from 0 (never), indicating not experiencing the symptom described in the item during the past week, to 3 (always), consistently experiencing the symptom. Total scores range from 0 to 30. A total score is calculated by summing the individual item scores. Higher scores indicate more severe depression. Here raw scores are reported. Population: This measure is only for 12-17 year olds, so only people in this age range are analysed. Initially, we enrolled 29 participants out of which 11 were 12-17 years old (analysed in first row). As we were interested in changes before and after the intervention, we also report the baseline results just for the participants who completed the outcome assessment. Out of the 15 participants who completed the outcome assessment, 7 were 12-17 years old (analysed in second row).
  units on a scale
    All Baseline Participants: number analyzed (Participants) | 11
    All Baseline Participants | 20 [17.5 to 23]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 7
    Participants who completed the Outcome Assessment | 18 [14.5 to 20.5]
Depression, Anxiety and Stress Scale (DASS-21) - Depression subscale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Depression subscale (7-items). Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), not experiencing depression symptoms during the past week to 3 (applied to me very much, or most of the time), frequently experiencing depression symptoms. Total scores range from 0 to 21. A total score is calculated by summing the individual item scores and then multiplying it by 2. Higher scores indicate more severe depression. Population: This measure is only for 18-25 year olds, so only people in this age range are analysed. Initially, we enrolled 29 participants out of which 18 were 18-25 years old (analysed in first row). As we were interested in changes before and after the intervention, we also report the baseline results just for the participants who completed the outcome assessment. Out of the 15 participants who completed the outcome assessment, 8 were 18-25 years old (analysed in second row).
  units on a scale
    All Baseline Participants: number analyzed (Participants) | 18
    All Baseline Participants | 35 [24.5 to 39.5]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 8
    Participants who completed the Outcome Assessment | 36 [35.5 to 40]
Depression, Anxiety and Stress Scale (DASS-21) - Anxiety subscale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Anxiety subscale (7-items). Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), not experiencing anxiety symptoms during the past week to 3 (applied to me very much, or most of the time), frequently experiencing anxiety symptoms. Total scores range from 0 to 21. A total score is calculated by summing the individual item scores and then multiplying it by 2. Higher scores indicate more severe anxiety. Population: This measure is only for 18-25 year olds, so only people in this age range are analysed. Initially, we enrolled 29 participants out of which 18 were 18-25 years old (analysed in first row). As we were interested in changes before and after the intervention, we also report the baseline results just for the participants who completed the outcome assessment. Out of the 15 participants who completed the outcome assessment, 8 were 18-25 years old (analysed in second row).
  units on a scale
    All Baseline Participants: number analyzed (Participants) | 18
    All Baseline Participants | 29 [18.5 to 36]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 8
    Participants who completed the Outcome Assessment | 36 [22.5 to 38.5]
Depression, Anxiety and Stress Scale (DASS-21) - Stress subscale [Median (Inter-Quartile Range); unit: units on a scale] — This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Stress subscale (7-items). Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), not experiencing stress symptoms during the past week to 3 (applied to me very much, or most of the time), frequently experiencing stress symptoms. Total scores range from 0 to 21. A total score is calculated by summing the individual item scores and then multiplying it by 2. Higher scores indicate more severe stress. Population: This measure is only for 18-25 year olds, so only people in this age range are analysed. Initially, we enrolled 29 participants out of which 18 were 18-25 years old (analysed in first row). As we were interested in changes before and after the intervention, we also report the baseline results just for the participants who completed the outcome assessment. Out of the 15 participants who completed the outcome assessment, 8 were 18-25 years old (analysed in second row).
  units on a scale
    All Baseline Participants: number analyzed (Participants) | 18
    All Baseline Participants | 35 [30 to 38]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 8
    Participants who completed the Outcome Assessment | 37 [33 to 38.5]
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) [Median (Inter-Quartile Range); unit: units on a scale] — This is a 14-item measure rated on a 5-point Likert scale, ranging from 1 to 5. A score of 1 ("none of the time"), indicates that the individual rarely or never experiences the feelings or behaviors described in the item, while a score of 5 ("all of the time") indicates that the individual frequently or always experiences these positive mental health states. The total score is calculated by summing the individual item scores, with possible scores ranging from 14 to 70, where higher scores indicate better mental well-being and a greater level of positive mental health. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 33 [28 to 39]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 32 [26 to 37.5]
Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Median (Inter-Quartile Range); unit: units on a scale] — This is an 18-item scale that measures general emotion regulation ability and various aspects of emotion regulation (in six subscales). Each item is rated on a 5-point Likert scale, with 1 ("Almost Never") indicating minimal difficulty with emotion regulation, and 5 ("Almost Always") indicating frequent or almost constant difficulty. The total score is calculated by summing the item scores ranging from 18 to 90. Higher scores indicate greater difficulty in regulating emotions. Conversely, lower scores suggest better emotion regulation skills. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 65 [58 to 69]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 66 [57.5 to 70]
11-item behaviour supplement to the Borderline Symptom List [Median (Inter-Quartile Range); unit: units on a scale] — This is an 11-item scale measuring engagement in other risky, self-destructive behaviours commonly associated with borderline personality disorder. Each item is rated on a Likert scale from 0 ("Not at all") indicating no engagement in the behavior during the assessed period, to 4 ("Daily or more often") indicating the participant engaged in the behavior on a daily basis or more frequently. Total scores are calculated by summing items and range from 0 to 44, with higher scores indicating more frequent or severe engagement in these behaviors. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 9 [6 to 12]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 10 [7 to 11.5]
Alcohol Use Disorders Identification Test (AUDIT) [Median (Inter-Quartile Range); unit: units on a scale] — This is a 10-item measure of alcohol misuse and possible dependence. Each item is rated on a 5-point scale ranging from 0 ("Never") not engaging in the behavior to 4 represents ("Daily or almost daily") highest level of engagement. The total score is obtained by summing the individual item scores, with the scale ranging from 0 to 40. Higher scores indicate a greater risk of alcohol misuse, with scores of 8 or higher commonly used to identify individuals at risk for hazardous or harmful drinking. Conversely, lower scores suggest minimal or no alcohol-related problems. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 6 [0 to 14]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 3 [0.5 to 11.5]
Cannabis Use Disorder Identification Test Revised (CUDIT-R) [Median (Inter-Quartile Range); unit: units on a scale] — Thisis an 8-item measure used to screen for problem cannabis use. Each item is rated on a 5-point Likert scale, where 0 ("Never") represents no engagement in the behavior, and 4 ("Daily or almost daily") represents the highest level of cannabis use. The total score is calculated by summing the responses, with the scale ranging from 0 to 40. A higher score indicates greater severity of cannabis misuse, and individuals with higher scores may be at risk for problematic cannabis use. Conversely, a lower score suggests minimal or no problematic cannabis use. Population: There was higher-than-expected attrition during the study. While we initially enrolled 29 participants (analysed in first row), only 15 completed the outcome assessment after the intervention duration. Therefore, as we were interested in changes before and after the intervention, we also report the baseline results for just the 15 participants who completed both baseline and outcome assessments (analysed in second row).
  units on a scale
    All Baseline Participants | 0 [0 to 1]
    Participants who completed the Outcome Assessment: number analyzed (Participants) | 15
    Participants who completed the Outcome Assessment | 0 [0 to 1.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Lost to Attrition
Description: Percentage of eligible enrolled participants not completing outcome assessment
Time Frame: 1 year
Population: 29 participants completed baseline assessment. Out of the 29, 14 did not complete the outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 29
Participants | 14

2. Primary Outcome: Number of Patients Adhering to Treatment
Description: Percentage of participants completing number of sessions as per-protocol (five sessions) out of the 27 participants who started therapy.
Time Frame: 3 months
Population: 29 eligible participants completed the baseline assessment. Out of the 29, 27 started therapy and 16 completed therapy per protocol meaning 3 face-to-face sessions and 2 follow up phone calls.
Measure: Count of Participants; unit: Participants
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 27
Participants | 16

3. Primary Outcome: User Experience Questionnaire
Description: This is an acceptability measure of app use designed to assess perceptions of the app, with items rated on a 7-point Likert scale ranging from -3 to +3. A score of -3 reflects the poorest user experience, while a score of +3 represents the highest level of satisfaction. A score of 0 indicates a neutral experience. The questionnaire consists of 26 items divided across six subscales: Attractiveness (overall impression), Perspicuity (ease of understanding), Efficiency (task completion speed), Dependability (reliability), Stimulation (engagement and enjoyment), and Novelty (innovation and creativity). For each of the six dimensions, the mean score of the items that correspond to that dimension is calculated. Higher scores across these subscales reflect a better overall user experience, while lower scores highlight specific areas for improvement. For the purposes of this analysis, the average of all dimensions mean scores were calculated for each participant.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 0.65 [0.27 to 1.28]

4. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: This is an 8 item version (Attkisson & Zwick, 1982) designed to provide a sensitive and comprehensive assessment of patient satisfaction with the therapy received. This was only administered post-treatment and sum scores were calculated for each participant. Each item is rated on a 4-point Likert scale, where responses range from 1 (very dissatisfied) to 4 (very satisfied). The individual scores from each item are summed to produce a total score for each participant, with a possible range of 8 (indicating low satisfaction) to 32 (indicating high satisfaction). Higher scores on the CSQ reflect greater overall satisfaction with the therapy received.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 25 [22 to 27.5]

5. Secondary Outcome: Timeline Follow-Back Technique (TLFB)
Description: This is an interview method conducted by the researcher who reconstructs together with the participant the number of self-harm behaviours using calendar cues. The scale records the total number of self-harm episodes within a specified timeframe of the last 3 months, with higher values indicating more frequent self-harm behaviours. The minimum number of episodes is 0 and the maximum number of episodes that can be reported for the 3 months is every day (so around 90 depending on the number of days of the month).
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
units on a scale | 0 [0 to 7]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — We used Wilcoxon Signed-Rank Test for our non-normally distributed data to compare scores before and after the Imaginator intervention; p = 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Self-Harm Imagery Interview (PANAS+)
Description: This interview is about mental images that deal with self-harm or occur with self-harm. It asks participants to think about one of these and explores their thoughts and emotions in relation to the image. This measure specifically assesses positive emotions on a 10-item scale. Each item is rated on a 5-point Likert scale with responses ranging from 1 (not at all), very low intensity or absence of the specific emotion, to 5 (extremely), extremely high intensity of that emotion. Scores range from 10 to 50, where a score of 10 reflects low positive emotional intensity, indicating weak or minimal positive emotions associated with the imagery, while a score of 50 represents high positive emotional intensity, signifying strong and vivid positive emotions. Higher scores indicate a greater intensity of positive emotional experiences related to the imagery.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 16 [13 to 18]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Self-Harm Imagery Interview (PANAS-)
Description: This interview is about mental images that deal with self-harm or occur with self-harm. It asks participants to think about one of these and explores their thoughts and emotions in relation to the image. This measure specifically assesses negative emotions on a 10-item scale. Each item is rated on a 5-point Likert scale with responses ranging from 1 (not at all), no negative emotional intensity, to 5 (extremely), extremely high negative emotional intensity. Scores range from 10 to 50, where a score of 10 reflects low negative emotional intensity, indicating weak or minimal negative emotions associated with the imagery, while a score of 50 represents high negative emotional intensity, signifying strong and intense negative emotions. Higher scores indicate a greater intensity of negative emotional experiences related to the imagery.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 36 [30 to 40.5]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: State Motivation for Reducing Self-harm (SM-SH) Scale
Description: This scale measures participants' motivation to control their self-harm through 12 items that measure the strength of their motivational cognitions in the present moment. Each item is rated on a 10-point Likert scale, ranging from 0 (never), indicating that the participant has no motivation or desire to control their self-harm at that moment, to 10 (constantly), , indicating that the participant has an extremely strong and persistent motivation to control their self-harm at that moment. Average scores are calculated for each participant ranging from 0 to 10, with higher scores indicating stronger motivation to control self-harm. This scale provides a sensitive measure of participants' current motivational state regarding self-harm reduction.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 6.33 [5.21 to 7.33]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Craving Experience Questionnaire for Self-Harm (CEQ-SH)
Description: This questionnaire assesses the urge to self-harm and assesses frequency, intensity, salience or dismissability of intrusive thoughts surrounding self-harm. It consists of 9 items, each rated on a 10-point Likert scale, ranging from 0 (not at all), indicating that the participant has no urge to self-harm or does not experience any intrusive thoughts related to self-harm, to 10 (constantly), indicating that the participant experiences a very strong and persistent urge to self-harm or is constantly preoccupied with thoughts of self-harm. The minimum score is 0, indicating no urge to self-harm, and the maximum score is 90, indicating the highest possible urge to self-harm. Higher scores reflect a stronger and more persistent urge to engage in self-harming behaviour.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 40 [21.5 to 50.5]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: Revised Children's Anxiety and Depression Scale (RCADS) - Anxiety Subscale
Description: This is a 47 item measure for 12-17 year olds with six sub-scales (separation anxiety disorder, social phobia, generalised anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder)). This analysis focuses on the Anxiety sub-scales (37 items), which consist of Separation Anxiety Disorder, Social Phobia, Generalised Anxiety Disorder, Panic Disorder, and Obsessive-Compulsive Disorder. Each item is scored from 0 (never), indicating not experiencing the symptom described in the item during the past week, to 3 (always), consistently experiencing the symptom. Total scores range from 0 to 111. A total score is calculated by summing the individual item scores. Higher scores indicate more severe anxiety. Here raw scores are reported.
Time Frame: 3 months
Population: Out of the 15 participants who completed the outcome assessment after the intervention, 7 were 12-17 years old.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 7
units on a scale | 49 [40.75 to 52]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

11. Other Pre Specified Outcome: Revised Children's Anxiety and Depression Scale (RCADS) - Depression Subscale
Description: This is a 47 item measure for 12-17 year olds with six sub-scales (separation anxiety disorder, social phobia, generalised anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder)). This analysis specifically focuses on the Depression subscale (10 items). Each item is scored from 0 (never), indicating not experiencing the symptom described in the item during the past week, to 3 (always), consistently experiencing the symptom. Total scores range from 0 to 30. A total score is calculated by summing the individual item scores. Higher scores indicate more severe depression. Here raw scores are reported.
Time Frame: 3 months
Population: Out of the 15 participants who completed the outcome assessment after the intervention, 7 were 12-17 years old.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 7
units on a scale | 14.5 [12 to 17.75]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

12. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (DASS-21) - Depression Subscale
Description: This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Depression subscale, which assesses symptoms associated with dysphoric mood, such as feelings of worthlessness. Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), indicating that the individual did not experience depression symptoms during the past week to 3 (applied to me very much, or most of the time), indicating that the individual frequently experienced depression symptoms. The Depression subscale consists of 7 items, with scores ranging from 0 to 21. Since the DASS-21 is a short version of the full scale, the total score for the Depression subscale is calculated by summing the individual item scores and then multiplying the final score by 2. Higher scores on this subscale indicate more severe depression, reflecting a higher intensity of depressive symptoms in the past week.
Time Frame: 3 months
Population: Out of the 15 participants who completed the outcome assessment after the intervention, 8 were 18-25 years old.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 8
score on a scale | 34 [20 to 36.5]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

13. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (DASS-21) - Anxiety Subscale
Description: This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Anxiety subscale, which measures symptoms associated with physiological arousal (e.g., trembling). Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), indicating that the individual did not experience anxiety symptoms during the past week to 3 (applied to me very much, or most of the time), indicating that the individual frequently experienced anxiety symptoms. The Anxiety subscale includes 7 items, with scores ranging from 0 to 21. Since the DASS-21 is a short version of the full scale, the total score for the Anxiety subscale is calculated by summing the individual item scores and multiplying the final score by 2. Higher scores on this subscale indicate more severe anxiety, reflecting greater physiological arousal and anxiety symptoms experienced over the past week.
Time Frame: 3 months
Population: Out of the 15 participants who completed the outcome assessment after the intervention, 8 were 18-25 years old.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 8
score on a scale | 22 [18 to 26]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

14. Other Pre Specified Outcome: Depression, Anxiety and Stress Scale (DASS-21) - Stress Subscale
Description: This is a 21-item scale for 18-25 year olds measuring levels of depression, anxiety and stress over the past week. This analysis focuses on the Stress subscale, which measures symptoms of tension and reactivity to stressful events. Each item is rated on a 4-point Likert scale, ranging from 0 (did not apply to me at all), indicating that the individual did not experience stress symptoms during the past week to 3 (applied to me very much, or most of the time), indicating that the individual frequently experienced stress symptoms. The Stress subscale includes 7 items, with scores for this subscale ranging from 0 to 21. Since the DASS-21 is a short version of the full scale, the total score for the Stress subscale is calculated by summing the individual item scores and multiplying the final score by 2 to adjust for the reduced number of items. Higher scores on this subscale indicate more severe stress, reflecting greater tension and reactivity to stressors over the past week.
Time Frame: 3 months
Population: Out of the 15 participants who completed the outcome assessment after the intervention, 8 were 18-25 years old.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 8
score on a scale | 28 [25.5 to 32.5]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

15. Other Pre Specified Outcome: Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
Description: This is a 14-item measure with positively worded items rated on a 5-point Likert scale, ranging from 1 to 5. A score of 1 ("none of the time") represents the lowest level of mental well-being, indicating that the individual rarely or never experiences the feelings or behaviors described in the item (e.g., feeling happy, confident, or connected). Conversely, a score of 5 ("all of the time") indicates the highest level of mental well-being, suggesting that the individual frequently or always experiences these positive mental health states. The total score is calculated by summing the individual item scores, with possible scores ranging from 14 to 70, where higher scores indicate better mental well-being and a greater level of positive mental health.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 41 [35.75 to 45]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

16. Other Pre Specified Outcome: Difficulties in Emotion Regulation Scale-Short Form (DERS-SF)
Description: This is an 18-item scale adapted from the original long version that measures general emotion regulation ability as well as various aspects of emotion regulation (in six subscales), e.g. difficulties engaging in goal directed behaviour when upset, and limited access to emotion regulation strategies. Each item is rated on a 5-point Likert scale, with 1 representing "Almost Never" (0-10% of the time), indicating minimal difficulty with emotion regulation, and 5 representing "Almost Always" (91-100% of the time), indicating frequent or almost constant difficulty. The total score is calculated by summing the item scores. The scale has a minimum value of 18 and a maximum value of 90. Higher scores indicate greater emotion regulation difficulties, reflecting more significant challenges in managing and regulating emotions. Conversely, lower scores suggest better emotion regulation skills and fewer difficulties in handling emotional responses.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 55.5 [51.25 to 63.5]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

17. Other Pre Specified Outcome: 11-item Behaviour Supplement to the Borderline Symptom List
Description: This is an 11-item scale measuring engagement in other risky, self-destructive behaviours (e.g., binge eating, substance misuse). The items are designed to assess the frequency and severity of these behaviors, which are commonly associated with borderline personality disorder. Each item is rated on a Likert scale from 0 to 4, with 0 representing "Not at all", indicating no engagement in the behavior during the assessed period, and 4 representing "Daily or more often", indicating the participant engaged in the behavior on a daily basis or more frequently. The total score is calculated by summing the responses. The scale has a minimum value of 0 and a maximum value of 44, with higher scores indicating more frequent or severe engagement in these behaviors.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 10 [4.25 to 11]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

18. Other Pre Specified Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: This is a 10-item measure of alcohol misuse and possible dependence, in which participants are asked to rate items related to their drinking (e.g. 'How often do you have a drink containing alcohol') on a 5-point scale ranging from 0 to 4. A score of 0 indicates "Never" engaging in the behavior (e.g., never drinking alcohol or never experiencing a specific consequence), while a score of 4 represents "Daily or almost daily", reflecting the highest level of engagement. The AUDIT is an effective means of identifying hazardous or harmful drinking behaviour. The total score is obtained by summing the individual item scores, with the scale ranging from 0 to 40. Higher scores indicate a greater risk of alcohol misuse, with scores of 8 or higher commonly used to identify individuals at risk for hazardous or harmful drinking. Conversely, lower scores suggest minimal or no alcohol-related problems.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 1 [0 to 4]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

19. Other Pre Specified Outcome: Cannabis Use Disorder Identification Test Revised (CUDIT-R)
Description: Thisis an 8-item measure used to screen for problem cannabis use. Participants are asked to rate a series of items related to their cannabis use (e.g., "How often do you use cannabis") on a 5-point Likert scale, where 0 represents "Never" or no engagement in the behavior, and 4 represents "Daily or almost daily", indicating the highest level of cannabis use. The total score is calculated by summing the responses, with the scale ranging from 0 to 40. A higher score indicates greater severity of cannabis misuse, and individuals with higher scores may be at risk for problematic cannabis use. Conversely, a lower score suggests minimal or no problematic cannabis use.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Imaginator App Plus Therapy
Number analyzed (Participants) | 15
score on a scale | 0 [0 to 0]
Statistical Analysis 1: Comparison: Imaginator App Plus Therapy; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The study run for 1 year and 2 months. Each participant completed the baseline assessment and waited on average 4.1 weeks (range 0.7 - 9) to start the intervention, while the average intervention duration was 21.3 weeks (range: 9.7 - 36). The outcome assessment would be conducted a week after completion of the intervention. Overall, each participant was assessed for approximately 6.5 months.
Description: To assess risk and adverse events, at the beginning of each session the therapist conducted the Columbia-Suicide Severity Rating Scale (C-SSRS) interview. Safety of the intervention determined by reviewing adverse events recorded at each assessment and therapy session/phone call contact
Arm/Group | Imaginator App Plus Therapy
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT06311084/Prot_SAP_001.pdf